CLINICAL TRIAL: NCT03033186
Title: Foreseeing the Moments of Occurrence of Everolimus Long-term Side Effects by Follow up of Trough Blood Concentrations
Brief Title: Everolimus TDM to Predict Long Term Toxicity
Acronym: Foresight
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL58486.068.16
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer; Renal Cell Carcinoma; Pancreatic Neuroendocrine Tumour; Gastrointestinal Neuroendocrine Tumour; Neuroendocrine Neoplasm of Lung
Keywords: Everolimus; Long term site effects; Dried Blood Spot; Therapeutic Drug Monitoring
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Renal Cell; Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and drop of blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Everolimus (afinitor): Patients using everolimus as therapy for cancer: Advanced (Hormone-Receptor [HR]-positive, HER2-negative) breast cancer (BC), advanced or unresectable neuroendocrine tumours of pancreatic (pNET), gastrointestinal or lung origin and metastatic renal cell carcinoma (mRCC)

SUMMARY:
Metastatic (HR-positive, HER2-negative) breast cancer (BC), advanced or unresectable neuroendocrine tumours of pancreatic (pNET), gastrointestinal or lung origin and metastatic renal cell carcinoma (mRCC) are diseases with poor outcome. Everolimus increases patients' median progression-free survival (PFS) with 4.6 months in metastatic BC (mBC), 7 months in (p)NET and 3 months in mRCC. However, serious adverse events (AEs) occur frequently. This reduces effectiveness of everolimus, because AEs are managed with dose reductions, treatment interruptions or even complete discontinuation of everolimus.

Therapeutic-drug-monitoring (TDM) is used to adjust the prescribed daily dose, to maintain effective everolimus whole blood concentrations, with the lowest possible risk of AEs. While everolimus TDM has been common in transplantation medicine, it has not been implemented in oncology.

The importance of TDM in oncology is supported by previous research which showed that a 2-fold increased everolimus whole blood trough concentration was associated with a short-term risk of grade ≥ 3 pneumonitis, stomatitis and metabolic events. Moreover, an exposure-toxicity relationship of everolimus in patients with thyroid cancer was observed, since initial everolimus concentrations could be associated with early toxicity (< 12 weeks, e.g. stomatitis). However, the association between initial everolimus measurements and long-term AEs (≥12 weeks, e.g. pneumonitis, anorexia and anemia) of any grade and the need for everolimus dose reductions could not be made. Since levels ±>18 µg/L were associated with toxicity, the investigators assume that the upper therapeutic window of everolimus in the oncologic setting will be ±18 µg/L. Similarly, a tendency to improved PFS and overall survival was observed when Cmin in steady state was above 14.1 μg/L. This seems to be the lower limit of the therapeutic window.

Before consensus about the feasibility of everolimus TDM in the oncologic setting can be achieved, a number of questions (the knowledge gaps) need to be answered: 1. It is unknown whether everolimus whole blood trough levels (over time) predict long-term AEs. 2. The optimal concentration range for everolimus, with the treatment of mBC, mRCC, or (p)NET is unknown, especially the upper limit associated with toxicity. 3. It is unknown what everolimus concentration level is associated with the need for everolimus dose reductions.

DETAILED DESCRIPTION:
Everolimus is an oral inhibitor of mammalian target of rapamycin (mTOR), a key signal transduction molecule of the phosphatidylinositol 3-kinase/Akt pathway. This pathway, which regulates cellular growth, proliferation, metabolism, survival and angiogenesis, is frequently dysregulated in human cancers and thus is a rational target for anticancer therapy. Everolimus is currently approved by the European Medicines Agency (EMA) and U.S. Food and Drug administration (FDA) for the treatment of different solid malignancies.

Metastatic (Hormone-Receptor [HR]-positive, HER2-negative) breast cancer (BC), advanced or unresectable neuroendocrine tumours of pancreatic (pNET), gastrointestinal or lung origin and metastatic renal cell carcinoma (mRCC) are diseases with poor outcome. Everolimus is part of palliative treatment and increases patients' median progression-free survival (PFS) with 4.6 months in metastatic BC (mBC), 7 months in pNET and 3 months in mRCC. However, serious adverse events (AEs) occur frequently; stomatitis up to 67%, non-infectious pneumonitis (NIP) up to 15%. This reduces effectiveness of everolimus, because AEs are managed with dose reductions, treatment interruptions or even complete discontinuation of everolimus.

Everolimus shows a large inter-individual pharmacokinetic variation in whole blood concentrations, due to variability in oral drug availability, patient non-compliance (e.g. due to drug-related toxicity, forgetting and/or overuse), drug-drug interactions with co-medication and many other factors. Furthermore, variation in the population pharmacokinetics of everolimus is caused by everolimus' hematocrit effect. This effect is present at high everolimus concentrations in combination with low hematocrit values, which is likely to be the case in the oncologic population. High incidences of anemia in oncologic patients treated with everolimus have been described, respectively being 32.1% (CI=17.5-51.3%) for all-grade (grades 1-4) toxicities and 6.9% (95% CI=4.1-11.3%) for high-grade (grades 3-4) toxicities. Therefore, studies have recommended to correct the everolimus whole blood concentrations for hematocrit determination.

The very different whole blood concentrations between individuals can result in supratherapeutic or subtherapeutic exposure levels and consequently in over- or undertreatment, respectively. Despite the inter-patient variability in systemic exposure, everolimus is currently prescribed at a fixed dose. Given the narrow therapeutic index and a positive exposure-efficacy relationship, there is a rationale for pharmacokinetically guided dosing also known as therapeutic drug monitoring (TDM) of everolimus. Such an approach could theoretically contribute to a tailor-made everolimus treatment with improved therapeutic efficacy and decreased risk for toxicity. Since daily everolimus dosing demonstrates dose proportionality and linear pharmacokinetics, this seems to be easily applicable. Furthermore, requirements for dose reduction at physicians discretion can be supported when it is known at what everolimus trough level a dose reduction is recommended.

Therapeutic-drug-monitoring (TDM) (i.e. measurement of everolimus whole blood levels after venipuncture) is used to adjust the prescribed daily dose, to maintain effective everolimus whole blood concentrations, with the lowest possible risk of AEs. In addition, TDM is a useful tool for early detection of non-adherence, and might also be used to monitor the effects of drug-drug interactions and food effects. While TDM, according to international consensus, has been common in transplantation medicine for 10 years, it has not been implemented in oncology. The importance of TDM in oncology is, however, supported by previous research that showed a 2-fold increased trough concentration (Cmin) of everolimus whole blood with a short-term risk of grade ≥ 3 pulmonary events (relative risk [RR] 1.9; 95% CI 1.1-3.3], stomatitis events (RR 1.5; 95% CI 1.1-2.1) and metabolic events (RR 1.3 95% 1.0-1.7). Moreover, an exposure-toxicity relationship of everolimus in patients with thyroid cancer was observed, since initial everolimus concentrations could be associated with early toxicity (< 12 weeks), i.e. stomatitis. However, the association between initial everolimus measurements and long-term AEs (≥ 12 weeks, e.g. pneumonitis, anorexia and anemia) of any grade and the need for everolimus dose reductions could not be made. Since a trough concentration of approximately 18 µg/L was associated with toxicity, the investigators assume that the upper therapeutic window of everolimus in the oncologic setting will be ±18 µg/L. Therefore, an upper threshold of >18 µg/L was considered for this study.Similarly, a tendency to improved PFS and overall survival (OS) was noted when CminSS was above 14.1 μg/L. This might be the lower limit of the therapeutic window.

However, the following knowledge gaps exist: 1. It is unknown whether everolimus trough whole blood levels (over time) predict for long-term AEs (≥12 weeks, e.g. pneumonitis, anorexia and anemia). 2. The optimal concentration range for everolimus, for the treatment of mBC, mRCC, or (p)NET is unknown, especially the upper limit associated with toxicity. 3. It is unknown what everolimus concentration level is associated with the need for everolimus dose reductions.

In order to quantitate the outcome toxicity, the number of dose reductions can be investigated as this is the sum of all different toxicities experienced by patients and these are also the toxicities that lead to clinical action by the treating physician. Furthermore, especially all NCI-CTCAE v4.0 grade ≥2 are important, and special attention should be focused on AEs that are highly prevalent, objectively measurable, clinically relevant and/or untreatable. These AEs will be leading to dose reductions or discontinuation of therapy.

Dose individualization based on the measured drug concentration could theoretically result in less toxicity and more efficacy. Further studies are required to determine the clinical utility of TDM for everolimus in oncology settings. Determination of everolimus concentrations at the onset of severe AEs (dose interruptions or reductions) and disease progression may enable better understanding of pathophysiology, permitting dose reduction at the right moment rather than drug withdrawal in patients with high everolimus concentrations. The clinical impact of this approach can be large, since everolimus treatment optimization is better than unnecessary switching to the next line of palliative treatment in these oncologic patients. This is supported by the study by Generali et al., finding the combination of everolimus plus exemestaan as first- or second-line therapy for mBC patients more efficacious than several chemotherapy regimens that were reported in the literature. Furthermore, it is important to realise that the initial concentration (< 12 weeks) does not reflect a change in steady-state trough concentration over time (≥12 weeks) due to various reasons. Some of them being drug-drug interactions, high-fat food effects, a change in haematocrit, non-adherence, dose-reductions and interruptions of the everolimus treatment.

Follow up of the everolimus concentration over time implies frequent pharmacokinetic sampling (blood draws). Nowadays everolimus exposure is determined by everolimus concentration measurement in whole blood. Therefore, a venipuncture is always necessary. This is invasive and requires patients to come to the hospital. It would be convenient for patients to have their everolimus concentration determined by dried blood spot (DBS) analysis. With DBS only a single drop of blood from the finger is necessary, which can be done at home and send by regular mail for analysis. Previous studies have showed the feasibility of the DBS approach in the oncologic setting. The physician may benefit from the ease of the DBS sampling method providing results timely before the patient visits the clinic for their (routine) check-up.

Previous methods for the measurement of everolimus by means of DBS have been developed. In the past, emphasis has been put on the development and analytical validation of the assay while the clinical validation was of minor importance. Some information has been gathered in transplantation medicine. However, in patients with cancer, the correlation between everolimus DBS concentrations and whole blood concentration is unknown. Furthermore, information regarding the important everolimus hematocrit effect in DBS at high concentration levels common in the oncology population is lacking. Therefore, the secondary objective is to determine the everolimus concentration collected with DBS from a finger prick and DBS paper spiked with a drop of venipunctured whole blood containing everolimus.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently treated with everolimus for any type of cancer, such as the EMA registered indications i.e. advanced (Hormone-Receptor [HR]-positive, HER2-negative) breast cancer, metastatic renal cell carcinoma (mRCC) or neuroendocrine tumour (NET) of pancreatic, gastrointestinal or lung origin.
* Aged 18 or above
* Able and willing to sign the informed consent

Exclusion Criteria:

* No informed consent
* Alactasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients currently treated with everolimus for any type of cancer, such as the EMA registered indications i.e. advanced (Hormone-Receptor [HR]-positive, HER2-negative) breast cancer, metastatic renal cell carcinoma (mRCC) or neuroendocrine tumours of pancreatic (pNET), gastrointestinal or lung origin.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Everolimus TDM to predict long-term toxicity | Up to 2 year
  The difference in percentage of patients with a high everolimus trough level (i.e. > 18 ng/mL) experiencing NCI-CTCAE v4.0 grade 2, 3 or 4 late AEs (i.e. toxicity reported from ≥ 12 weeks onward, e.g. pneumonitis, anorexia, anemia) compared to participants with lower trough concentrations.

SECONDARY OUTCOMES:
Everolimus TDM to predict short-term toxicity | Up to 2 year
  The difference in percentage of patients with a high everolimus trough level (i.e. > 18 ng/mL) experiencing NCI-CTCAE v4.0 grade 2, 3 or 4 early AEs (i.e. toxicity reported from < 12 weeks, e.g. stomatitis) compared to participants with lower trough concentrations.
Correlation everolimus concentration DBS from fingerprick with whole blood from venipuncture | Up to 2 year
  To define the correlation between everolimus concentration measured in whole blood after a venipuncture as compared to the everolimus concentration measured from dried capillary blood extracted from the Whatman filterpaper of the DBS.
Correlation everolimus concentration DBS from fingerprick with DBS spiked with whole blood from venipuncture | Up to 2 year
  To define the correlation between everolimus concentration collected with DBS from a finger prick and DBS paper spiked with a drop of everolimus from venipunctured whole blood extracted from the Whatman filterpaper of the DBS.
Everolimus TDM to predict dose reductions | Up to 2 year
  To define the correlation between the everolimus trough levels (over time) between patients using full dose everolimus (e.g. 10 mg once daily) and patients using everolimus in a reduced dose (e.g. 2,5 or 5 mg once daily) at each moment of blood sampling in time.

CONTACTS AND LOCATIONS:
Overall Officials: S. Croes, PharmD, PhD, Principal Investigator — Maastricht University Medical Centre+
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No